CLINICAL TRIAL: NCT03607877
Title: Gender Differences and Influence of Walking Exercise and a Psychosocial Intervention on Psychological Well-being and Sense of Coherence Amongst Retried Senior Citizens
Brief Title: A RCT of Walking With Positive Education in Retired Elders
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Hui-Hsun Chiang, Assistant Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Exercise and Psychology
Record Dates: First submitted 2018-07-13; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Happiness; Educational Problems; Exercise
Keywords: Positive education; Walking exercise; Well-being; Pedometer; Cardiovascular fitness
MeSH Terms: conditions — Motor Activity | interventions — Walking

STUDY DESIGN:
Intervention Model Description: Three arms of experimental design were used: Pedometer walking training (PWT), positive education and pedometer walking training (PEPWT), and pedometer walking (PW). Trained walking exercise was provided by a physical education expert three times per week, 45 minutes per session. Positive education was designed and led by a licensed psychologist. Six sessions of activities targeted participants' self-strength, competence and self-efficacy in walking exercise; positive relations with others; and positive emotions about life and healthy lifestyle. Of 150 participants, 60, 60 and 30 were randomly assigned to PWT, PEPWT, and PW, respectively. Demographic information, Chinese Happiness Inventory (CHI), regular walking exercise and six-minute walking distance were assessed before and after the intervention.
Who Masked: Investigator
Masking Description: Randomization was conducted using opaque envelops and a randomly generated number sequence by an independent research assistant who had no prior knowledge of the recruited elders. Researchers allocated participants to their treatment condition based on the randomization code in the sealed envelope (opened in order of sequence). Investigator was blind to participants, but researchers were not blind to the patients' treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pedometer walking (PW) (Active Comparator): 15 minutes of warm-up activities, 30 minutes of walking, and 10 minutes to cool down for 3 months.
  Interventions: Behavioral: pedometer walking
- pedometer walking with training (PWT) (Active Comparator): 15 minutes of warm-up activities, 30 minutes of walking, and 10 minutes to cool down. Exercise intensity for the first four weeks was 50-55% heart rate reserve (HRR) with training for 3 months.
  Interventions: Behavioral: Pedometer walking with training
- positive education and walking (PEPWT) (Experimental): PEPWT: 15 minutes of warm-up activities, 30 minutes of walking, and 10 minutes to cool down for 3 months and six sessions of positive education.
  Interventions: Behavioral: Pedometer walking training and positive education

INTERVENTIONS:
Behavioral: Pedometer walking training and positive education — Intervention: (1)Positive education: Six psychosocial sessions were designed to enhance elders' positive emotion, motivation and self-efficacy to walk.
  (2) Pedometer walking training: walk at least 30 minutes per day and at least three times per week with family support and exercise companions.
  Other Names: walking exercise
  Arms: positive education and walking (PEPWT)
Behavioral: Pedometer walking with training — Intervention:walk at least 30 minutes per day and at least three times per week with family support and exercise companions.
  Other Names: walking exercise
  Arms: pedometer walking with training (PWT)
Behavioral: pedometer walking — Intervention: pedometer walking at least 30 minutes per day and at least three times per week
  Other Names: walking
  Arms: pedometer walking (PW)

SUMMARY:
Three arms of experimental design were used: Pedometer walking training (PWT), positive education and pedometer walking training (PEPWT), and pedometer walking (PW). Trained walking exercise was provided by a physical education expert three times per week, 45 minutes per session. Positive education was designed and led by a licensed psychologist. Six sessions of activities targeted participants' self-strength, competence and self-efficacy in walking exercise; positive relations with others; and positive emotions about life and healthy lifestyle. Of 150 participants, 60, 60 and 30 were randomly assigned to PWT, PEPWT, and PW, respectively. Demographic information, Chinese Happiness Inventory (CHI), regular walking exercise and six-minute walking distance were assessed before and after the intervention.

DETAILED DESCRIPTION:
Randomization (allocation ratio 2:2:1) was stratified to three arms: pedometer walking (PW), pedometer walking with training (PWT), and positive education and pedometer walking with training (PEPWT). Randomization was conducted using opaque envelops and a randomly generated number sequence by an independent research assistant who had no prior knowledge of the recruited elders. Researchers allocated participants to their treatment condition based on the randomization code in the sealed envelope (opened in order of sequence). Researchers were not blind to the patients' treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria included being retired from work and being at least 55 years old.

Exclusion Criteria:

* Elders who had cardiovascular disease, who were unable to walk, who had dementia or psychiatric disease, who already exercised regularly, or who were unwilling to sign the consent form were excluded from the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2012-03-06 (Actual); Study Completion 2012-06-30 (Actual)

PRIMARY OUTCOMES:
Chinese Happiness Inventory | 3 months
  Chinese Happiness Inventory (CHI). The CHI 20-item version has been widely used to measure individual well-being in Chinese culture (Lu & Shih, 1997; Chiang, Lin, & Lee, 2016). Each statement represents a different level of happiness, ranging from 0 (very dissatisfied) to 3 (very satisfied). CHI score is the sum of 20 items. The higher the score is, the higher the psychological well-being is. CHI has high validity and reliability (Lu & Shih, 1997; Chiang, Lin, & Lee, 2016).
Cardiovascular fitness | 3 months
  Cardiovascular fitness was calculated by using the six-minute walk test (6MWT) which measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface and has been suggested as a useful outcome tool (Du, Newton, Salamonson, Carrieri-Kohlman, & Davidson, 2009). The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. The 6MWT has been used to detect changes following interventions to improve exercise tolerance for healthy older adults (Troosters, Gosselink, & Decramer, 1999).

CONTACTS AND LOCATIONS:
Overall Officials: Tony Szu-Hsien Lee, Prof, Principal Investigator — Health Education and Health Promotion, National Taiwan Normal University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Du H, Newton PJ, Salamonson Y, Carrieri-Kohlman VL, Davidson PM. A review of the six-minute walk test: its implication as a self-administered assessment tool. Eur J Cardiovasc Nurs. 2009 Mar;8(1):2-8. doi: 10.1016/j.ejcnurse.2008.07.001. Epub 2008 Aug 9. PMID 18694656
- See also: Meta-analysis — https://www.ncbi.nlm.nih.gov/pubmed/18694656